CLINICAL TRIAL: NCT06199271
Title: Neoadjuvant Adebrelimab Plus Dalpiciclib in HPV-negative Locally Advanced Head and Neck Squamous Cell Carcinoma: A Phase II Clinical Trial
Brief Title: Neoadjuvant Adebrelimab Plus Dalpiciclib in Head and Neck Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhongzheng Xiang (Other)
Responsible Party: Sponsor-Investigator, Zhongzheng Xiang, Research associate, Sichuan University
Organization: Sichuan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Neo-AdDa
Record Dates: First submitted 2023-12-01; First posted 2024-01-10 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Neoadjuvant therapy; Immunotherapy; CDK4/6 inhibitor; Locally advanced head and neck squamous cell carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — dalpiciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Patients with resectable locally advanced head and neck squamous carcinoma cell carcinoma receive adebrelimab plus dalpiciclib before surgery.
  Interventions: Drug: Adebrelimab and dalpiciclib

INTERVENTIONS:
Drug: Adebrelimab and dalpiciclib — Before surgery, the eligible patients received 3 cycles of adebrelimab (1200 mg intravenously every 3 weeks, Day 1, 22 and 43) and 2 cycles of dalpiciclib (150 mg, po, every 4 weeks, day 1-21 and 29-49). Administration dose adjustments were permitted according to the haematological or non-haematological toxicity.
  Other Names: Dalpiclib hydroxyethanesulfonate tablets; Adebrelimab iniection

SUMMARY:
This study is a single arm phase II trial including 30 patients with III-IVB (according to the 8th edition of UICC/AJCC staging) locally advanced head and neck squamous cell carcinoma (HNSCC) eligible for resection, who receive Adebrelimab plus Dalpiciclib as neoadjuvant regimen before surgery.

This proposed study will evaluate the efficacy and safety of preoperative administration of Adebrelimab plus Dalpiciclib in HNSCC who are eligible for resection.

DETAILED DESCRIPTION:
In this study, eligible patients will be enrolled into study arm to accept study treatment. Pathological response rate and objective response rate will be the primary outcome measures. Adverse events will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically diagnosed with HPV-negative head and neck squamous cell carcinoma (HNSCC), including oral, laryngeal, hypopharyngeal, and HPV-negative oropharyngeal carcinoma (with HPV testing methods for oropharyngeal carcinoma, including p16 immunohistochemistry or HPV DNA tests).
2. Patients with resectable locally advanced head and neck squamous cell carcinoma (LA-HNSCC), classified as stage III-IVB according to the 8th edition of UICC/AJCC staging.
3. Age greater than or equal to 18 and less than 75 at the time of study entry.
4. Karnofsky Performance Status (KPS) score ≥ 70 points.
5. No prior exposure to other relevant anti-tumor treatments.
6. No distant metastasis (DM).
7. Intention to undergo curative treatment.
8. Adequate bone marrow function: total white blood cell count ≥ 3.5 × 10^9 /L, absolute lymphocyte count ≥ 0.8 × 10^9/L, absolute neutrophil count ≥ 1.5 × 10^9/L, platelets ≥ 100 × 10^9 /L, hemoglobin ≥ 90g/L.
9. Adequate hepatic function: bilirubin ≤ 1.5 x ULN; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN.
10. Adequate renal function: serum creatinine ≤ 1.5 x ULN, creatinine clearance (Ccr) ≥ 60 ml/min (if using the Cockcroft-Gault formula), urinalysis indicating urinary protein less than 2+, or 24-hour urinary protein quantification < 1g.
11. Adequate coagulation function: international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 x ULN. If the subject is currently receiving anticoagulant therapy, PT within the therapeutic range of the anticoagulant can be accepted.
12. No severe organic heart disease and arrhythmia.
13. Women of childbearing age (15-49 years) must have a negative pregnancy test within 7 days before treatment. Both men and women of reproductive age must use highly effective contraception during the study and for 3 months after treatment.
14. Willingness and ability to sign an approved Informed Consent Form.

Exclusion Criteria:

1. Previous treatment of any other form of anti-tumor therapy;
2. Patients with allergies and congenital immunodeficiency;
3. active infection;
4. Previous organ transplantation;
5. History of autoimmune diseases or other conditions requiring prolonged systemic use of corticosteroids or immunosuppressive therapy;
6. Patients with a history of use of the following drugs (CYP3A4 inhibitors: clarithromycin, indinavir, itraconazole, ketoconazole, lopinavir, ritonavir, nefazodone, nelfinavir, posaconazole, saquinavir, telaprevir, telithromycin, voriconazole and grape sleeve or grape sleeve juice, ziprasidone, lorlostazol, ticagrelor, aprepitant, netupitant, ondansetron, domperidone, etc.; CYP3A4 inducers: rifampicin, carbamazepine, enzalutamide, phenytoin, rifampicin and St. John's wort, efaviren, bosentan, modafinil, etc.);
7. Human Immunodeficiency Virus (HIV) positive;
8. Active hepatitis B or C infection (HBV DNA, HCV RNA exceeding normal upper limits);
9. Abnormal blood counts: White blood cells <3.5×10^9/L, absolute lymphocyte count <0.8×10^9/L, neutrophils <1.5×10^9/L, platelets <100×10^9/L, hemoglobin <90g/L; elevated bilirubin >1.5 times the upper limit of normal, transaminases (AST, ALT) >3 times the upper limit of normal (5 times if liver metastasis), serum creatinine >1.5 times the upper limit of normal; abnormal coagulation function, international normalized ratio (INR) or prothrombin time (PT) >1.5 times the upper limit of normal.
10. Severe cardiovascular, respiratory, or immune system diseases, including urinary obstruction, positive cardiac stress test, myocardial infarction, arrhythmias, obstructive or restrictive lung disease, or other diseases that investigators believe may increase the risk of subjects.
11. Pregnant or lactating females;
12. Patients unwilling to use effective contraception during the treatment period and the following 3 months.
13. Simultaneous participation in other clinical studies.
14. Patients in critical condition unable to complete the investigation.
15. Patients with a history of mental illness (e.g., schizophrenia, bipolar disorder, anxiety disorders, depression, phobias, etc.) or those diagnosed with a mental disorder at the time of clinical trial enrollment or their spouses.
16. Patients or spouses experiencing communication barriers or inability to respond normally due to reasons such as confusion, aphasia, intellectual disability, etc.
17. Presence of other malignant tumor diseases.
18. Other factors deemed unsuitable or likely to affect the subject's participation or completion of the study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological response rate | 1-year
  The pathological response was evaluated by pTR (the appearance of tumor necrotic cells and keratin fragments with giant cell/tissue cell responses), including significant pathological response (Major pathological response, MPR, pTR-2 ≥ 50%), partial pathological response (Partial pathological response, PPR, pTR-1 10% -49%), and no pathological response (Non pathological response, NPR, pTR-0<10%).